CLINICAL TRIAL: NCT06683105
Title: A Pilot Randomized Trial Investigating the MyIBDDiet App to Improve Self-management of an Anti-inflammatory Diet for Individuals With Inflammatory Bowel Disease
Brief Title: Clinical Investigation of MYIBDDiet App Developed for Inflammatory Bowel Disease (IBD) Patients to Self-manage Their Diet
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00141681
Record Dates: First submitted 2024-11-05; First posted 2024-11-12 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Inflammatory Bowel Disease (IBD)
Keywords: Inflammatory Bowel Disease (IBD); Crohn's disease; Ulcerative colitis; Self-management; Malnutrition; Mediterranean diet; Mobile health applications
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative; Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator): This group will not use the app for the first 30 days, then begin using it for the following 30 days.
  Interventions: Other: MyIBDDiet app
- MyIBDDiet users (Experimental): This group will use the MyIBDDiet app for 60 days and compared with the standard of care group.
  Interventions: Other: MyIBDDiet app

INTERVENTIONS:
Other: MyIBDDiet app — Participants in the Standard of Care arm will be administered the intervention (using the app) for 30 days, and participants in the MYIBDDiet arm will use the app for 60 days.

SUMMARY:
The goal of this clinical trial is to learn if an app designed for diet education can help patients with inflammatory bowel disease (IBD) learn about healthy eating.

The main question[s] it aims to answer are:

* Is the app easy to use?
* Is the app useful? Researchers will compare the diet app to see if it is better at teaching patients about a healthy diet than the standard information they may receive from their doctor.

Participants will be asked to use the app for one month and answer surveys to see how easy the app is to use and if it leads to healthier eating.

DETAILED DESCRIPTION:
(Background): Inflammatory bowel disease (IBD), encompassing Crohn's disease and ulcerative colitis affects various segments of the gastrointestinal tract. Although this is a chronic illness, patients may experience periods of active inflammation and inactive disease or remission. At diagnosis, patients commonly enquire about what they should not be eating or avoiding. In the past, advice was limited to vague recommendations to "avoid the foods that bother participants" due to lack of research data to support a specific diet as beneficial.

The etiopathogenesis of IBD is thought to involves genetic predisposition, an altered composition and function of the intestinal microbiome, and a dysregulated immune. Diet has been shown to play a role in modulating the intestinal microbiome. There is now growing evidence to support the role of diet in in the management of IBD and recent guidelines have made more concrete recommendations for Mediterranean diet and avoidance of ultra-processed foods.

Although gastroenterologists may be aware and able to advice patients on the type of diet, few would have the expertise or time to provide specific details of the foods that are allowed or excluded in these diets. Not all patients will have access to a dietician and those who have access to a consultation will not have regular reinforcement of the concepts discussed.

The investigators therefore propose a digital solution to bridge the gap in care and allow for daily reinforcement of nutrition knowledge to help patients adhere to a healthy eating pattern. The MyIBDDiet app is designed to allow for tracking of food intake including preparation method, added fats and food processing with immediate messaging feedback on whether the food item should be consumed more often or less often. Symptom tracking will allow patients to correlate how they felt to their food intake. Additionally, further education and resources will be provided in the form of short videos or visual tools. These resources will be developed in response to user requests.

In this randomized pilot trial study, the investigators aim to conduct a clinical investigation to evaluate the effects of the the intervention of using the educational diet tracking app (MyIBDDiet).

(Purpose): The investigators aim to evaluate the MyIBDDiet app, designed to improve self-management of a healthy eating pattern.

(Hypothesis): It is hypothesized that diet plays a role in modulating the intestinal microbiome. A Western diet high in saturated fat, sugar and processed foods contributes to intestinal microbiome dysbiosis and has been implicated in the pathogenesis of IBD. Conversely, an anti-inflammatory pattern of eating (e.g., the Mediterranean diet) with concomitant reduction in processed foods has recently been cited by the American Gastroenterology Association as an adjunct to inactive states of IBD.

Majority (85.4%) of individuals living with IBD believe diet is implicated in disease relapse. A paucity of established dietary guidance has led patients with IBD to self-impose dietary restrictions, thus further increasing risk of malnutrition. Furthermore, while larger centers are more likely to be associated with dedicated nutrition professionals, most with IBD may be faced with navigating nutrition misinformation associated with random websites and the IBD community, itself.

(Justification): Mobile health applications (apps) providing self-managed, evidenced-based diet and lifestyle programs are emerging for the IBD population. While many IBD-related apps exist, some of the apps focus solely on tracking without providing education while others provide recipes or therapeutic diets that require coaching. Few focus on diet education or self-management. As such, the investigators aim to develop a nutrition app that delivers up-to-date, evidenced-based diet information in a format that follows principles of adult learning. Newly developed electronic resources and videos will provide education on an anti-inflammatory pattern of eating, fiber and the intestinal microbiome, food additives and emulsifiers and practical substitutions in a restaurant setting will be made available in the app. Our goal is to expand beyond surface learning (i.e. Videos/handouts) to try to achieve a deeper level of understanding by having patients categorize their food intake while tracking with immediate feedback on the rationale behind the recommendation to choose the item more or less often.

By integrating videos, tutorials, and patient entries, MyIBDDiet app combines clinical advice with patient independence, and empowerment.

(Objectives): The objectives include evaluating the safety and efficacy of the app in improving diet quality and diet knowledge.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years
2. Able to provide informed consent
3. Established diagnosis of IBD determined by treating physician
4. Not in acute flare
5. Not pregnant
6. Willing and able to comply with all required study procedures

Exclusion Criteria:

1. Short bowel syndrome
2. High ostomy output
3. Intestinal strictures
4. Pregnancy or breastfeeding
5. Malnutrition (evaluated by Canadian Nutrition Screening Tool (CNST) )
6. Conditions requiring dietary restrictions (e.g. Celiac disease, kidney disease, diabetes, eosinophilic esophagitis)
7. Have other conditions that may require low fibre diet such as irritable bowel syndrome, gastroparesis.
8. Currently on a therapeutic diet
9. Have ever participated in another therapeutic diet study
10. Already on a diet for IBD or using diet tool for IBD (e.g. Mediterranean or anti-inflammatory diet)
11. Active malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Diet quality | Through study completion, an average of 1 year
  Change in diet quality before and after using MyIBDDiet App assessed using the Mini-EAT tool and Healthy Eating Index (HEI)

SECONDARY OUTCOMES:
Quality of live | Through study completion, an average of 1 year
  Quality of life will be assessed by European Quality of Life Five Dimension (EQ-5D) questionnaire

OTHER OUTCOMES:
Change in adherence to / knowledge of Mediterranean diet | Through study completion, an average of 1 year
  Determined with Mediterranean Diet Serving Score (MDSS)
Change in intake of highly processed foods | Through study completion, an average of 1 year
  Change in intake of highly processed foods as determined by Automated Self-Administered 24-Hour Dietary Recall (ASA24®) (Dietary Assessment) Tool and NOVA classification. (NOVA classification groups foods according to the nature, extent and purpose of the industrial processing they undergo).

CONTACTS AND LOCATIONS:
Locations (1):
- Zeidler Ledcor Centre, University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gubatan J, Kulkarni CV, Talamantes SM, Temby M, Fardeen T, Sinha SR. Dietary Exposures and Interventions in Inflammatory Bowel Disease: Current Evidence and Emerging Concepts. Nutrients. 2023 Jan 22;15(3):579. doi: 10.3390/nu15030579. PMID 36771288
- [Result] Gold SL, Chiew BA, Rajagopalan V, Lavallee CM. Identification and Evaluation of Mobile Applications for Self-Management of Diet and Lifestyle for Patients with Inflammatory Bowel Disease. J Can Assoc Gastroenterol. 2023 Sep 16;6(5):186-195. doi: 10.1093/jcag/gwad029. eCollection 2023 Oct. PMID 37811532
- [Result] Godala M, Gaszynska E, Durko L, Malecka-Wojciesko E. Dietary Behaviors and Beliefs in Patients with Inflammatory Bowel Disease. J Clin Med. 2023 May 14;12(10):3455. doi: 10.3390/jcm12103455. PMID 37240560
- [Result] Sekhon M, Cartwright M, Francis JJ. Development of a theory-informed questionnaire to assess the acceptability of healthcare interventions. BMC Health Serv Res. 2022 Mar 1;22(1):279. doi: 10.1186/s12913-022-07577-3. PMID 35232455
- [Result] Balestrieri P, Ribolsi M, Guarino MPL, Emerenziani S, Altomare A, Cicala M. Nutritional Aspects in Inflammatory Bowel Diseases. Nutrients. 2020 Jan 31;12(2):372. doi: 10.3390/nu12020372. PMID 32023881
- See also: Related Info — https://asa24.nci.nih.gov/demo/
- See also: Related Info — https://redcap.ualberta.ca/